CLINICAL TRIAL: NCT04028310
Title: Developmental Dyslexia and Remediation Methods. Phonological, Visual-attentional and Cross-modal Approaches, a Multicentric Study.
Brief Title: Developmental Dyslexia and Remediation Methods
Acronym: DDMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 19-HPNCL-02
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Dyslexia, Developmental
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phonological group (Experimental)
  Interventions: Other: Phonological
- visual-attention group (Experimental)
  Interventions: Other: Visual-attention

INTERVENTIONS:
Other: Phonological — * Phase 1: intervention without targeted daily training (30 minutes/ week, for 8 weeks)
  * Phase 2: intervention with targeted daily training
    * Phonological training (15 minutes/ day, 5 days/week, for 8 weeks)
    * Visuo-attentional training (15 minutes/ day, 5 days/week, for 8 weeks)
    * Cross-modal training (15 minutes/ day, 5 days/week, for 8 weeks)
  * Phase 3: stopping training sessions for 8 weeks
  Arms: Phonological group
Other: Visual-attention — * Phase 1: intervention without targeted daily training (30 minutes/ week, for 8 weeks)
  * Phase 2: intervention with targeted daily training
    * Visuo-attentional training (15 minutes/ day, 5 days/week, for 8 weeks)
    * Phonological training (15 minutes/ day, 5 days/week, for 8 weeks)
    * Cross-modal training (15 minutes/ day, 5 days/week, for 8 weeks)
  * Phase 3: stopping training sessions for 8 weeks
  Arms: visual-attention group

SUMMARY:
At least, three theoretical frameworks are currently involved in therapeutic research in developmental dyslexia. Each theoretical framework relies on the type of underlying cognitive processes that is viewed as impaired: 1°) phonological processing, 2°) cross modal integration, 3°) visual attention processing. In this controlled and randomized study, three types of computerized training are combined in a multi-factorial remedial approach in 8 to 12 year old children with dyslexia. The main objective is to compare the effectiveness of this remedial approach which combines phonological, visual-attentional and cross-modal training with conventional non-intensive and non-specific rehabilitation

DETAILED DESCRIPTION:
Developmental dyslexia is defined as a specific and lasting reading learning disorder. This neurodevelopmental disorder has a severe impact on overall academic learning and behavior, compromises professional and social development and affects 10% of school-age children. As a public health problem, its diagnosis and management are still highly controversial, and the lack of scientific consensus leads to great heterogeneity in clinical practices and post-treatment outcomes. Three therapeutic axes guide research for developmental dyslexia. The first axis is based on phonological deficits. According to the phonological representation hypothesis, a specific deficit in the processing of phonological representations that support the identification of sounds is the cause of the reading disorder. The second axis focuses on attention-related cognitive deficits. According to the visuo-attention deficit hypothesis, a lack of the visuo-attention processing can be viewed as one of the explanatory causes of a dysfunction in letter identification and reading procedures. The third axis aims to achieve automatized processing for letter/sound association. According to the axis, a lack of cross-modal integration in word decoding is altered by a lack of simultaneous association between of a visual and an auditory stimulus.

Many studies attempted to exclusively validate selective remediation according to causal hypotheses that are mainly cross-modal, phonological or visuo-attentional. However, the evaluation of these underlying processing in dyslexic children shows great clinical heterogeneity since most of children simultaneously have the three deficits. Furthermore, no study evaluates the benefits of combining these different trainings on reading skills.

In this controlled and randomized study, three types of computerized training are combined in a multi-factorial remedial approach in 8 to 12 year old children with dyslexia. The main objective is to compare the effectiveness of this remedial approach which combines phonological, visual-attentional and cross-modal training with conventional non-intensive and non-specific rehabilitation.

The secondary objectives will be 1°) to compare the effectiveness on reading skills of a phonological training, versus a visuo-attentional training, 2°) to compare the effectiveness on reading skills from in the order of phonological and visuo-attentional training, 3°) to compare the evolution of performance in comprehension and written production at the end of the three training sessions and 4°) to evaluate child and parents' perception for the outcome of the reading disorder at the end of the training sessions using Likert scales, by means of a questionnaire. The analysis of the results will make possible to evaluate a remedial approach to dyslexia in a clinical context and to better understanding and management of written language disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 years old and ≤ at 13 years old;
* Diagnosis of dyslexia validated by performances ≤ at -1.5 standard deviations from the mean on leximetric tests.
* Diagnosis of mixed dyslexia validated by performances ≤ at -1.5 standard deviations from the mean for reading irregular words and pseudo-words in the Evalec© test.
* Performance ≤ at -1.5 standard deviations from the mean for phonological (Evalec©) and visual-attentional tasks in the Evadys© and Sigl© tests.
* Home equipped with a connected computer system for daily training.
* Signing of informed consent by the parents
* The child must be affiliated to a social security scheme

Exclusion Criteria:

* Intellectual retardation, neurological disorders, pervasive developmental disorder;
* Primary sensory deficit;
* Educational deficiencies;
* attention deficit hyperactivity disorder, dysphasia;
* Previous daily phonological or visual-attentional training.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
reading skills effectiveness | 26 weeks to baseline
  measure of reading level (reading age) : accuracy (number of errors) and reading time (in seconds) in raw scores and standard deviation

SECONDARY OUTCOMES:
reading skills effectiveness 8 weeks | 8 weeks to baseline
  Measure of reading level : accuracy (error rates) and reading time (in milliseconds) in raw scores and standard deviations
reading skills effectiveness 18 weeks | 18 weeks to baseline
  Measure of reading level : accuracy (error rates) and reading time (in milliseconds) in raw scores and standard deviations
orthographic skills effectiveness | 26 weeks to baseline
  count of orthographic (number of errors) in raw scores and standard deviation
reading comprehension skills effectiveness | 26 weeks to baseline
  measure of reading comprehension level (error rates) in raw scores and standard deviation
perception of the evolution of the reading disorder | 26 weeks to baseline
  measure the perception of the evolution of the reading disorder by Likert scales : Number of items: 13
  * Score from 5 to 1
  * For example, "I like to read" a lot = 5, a lot = 4, normal" = 3, a little = 2, not at all = 1 Another example "it's easy to read", really very easy = 5, I do well = 4, normal = 3, a little difficult = 4, very difficult = 1
  * The maximum value 5 means that reading and learning are perceived very positively
  * The minimum value 1 means that reading and learning are perceived very negatively
  * Results: An increase in scores measured before and after the three training sessions means an improvement

CONTACTS AND LOCATIONS:
Overall Officials: HARRAR-ESKINAZI KARINE, Principal Investigator — CERTA Fondation Lenval, Children Hospital of Nice CHU-LENVAL
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France

REFERENCES:
- [Derived] Darrot G, Gros A, Manera V, De Cara B, Faure S, Corveleyn X, Harrar-Eskinazi K. Effects of a developmental dyslexia remediation protocol based on the training of audio-phonological cognitive processes in dyslexic children with high intellectual potential: study protocol for a multiple-baseline single-case experimental design. BMC Pediatr. 2023 Aug 17;23(1):404. doi: 10.1186/s12887-023-04189-6. PMID 37592217
- [Derived] Harrar-Eskinazi KL, De Cara B, Leloup G, Nothelier J, Caci H, Ziegler JC, Faure S. Multimodal intervention in 8- to 13-year-old French dyslexic readers: Study protocol for a randomized multicenter controlled crossover trial. BMC Pediatr. 2022 Dec 28;22(1):741. doi: 10.1186/s12887-022-03701-8. PMID 36578007